CLINICAL TRIAL: NCT00164216
Title: Evaluation of the Efficacy and Effectiveness of Combined Therapy With Mefloquine and Artesunate for Uncomplicated Malaria Treatment in the Loreto Region (Amazon Basin), Peru
Brief Title: Efficacy and Effectiveness of Combined Therapy for Uncomplicated Malaria Treatment in Peru
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: National Institute of Health, Peru (Other)
Responsible Party: Sponsor
Other Study IDs: CDC-NCID-4476
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Malaria Falciparum
Keywords: malaria; combination therapy; mefloquine; artesunate; Peru; malaria, uncomplicated
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Mefloquine; Artesunate

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: mefloquine plus artesunate

SUMMARY:
This is a study of the efficacy and effectiveness of combination therapy for malaria due to P. falciparum in the Loreto Department, Iquitos, Peru. The investigators will enroll subjects ≥ 1 year-old who have a diagnosis of uncomplicated malaria due to P. falciparum. Patients will receive a treatment regimen consisting of mefloquine (25 mg/kg per day for two days) and artesunate (12 mg/kg per day for three days). Patients will be divided into two groups: one will receive drugs under direct supervision and the other will be instructed on how to take the drugs by themselves. Clinical and parasitologic response will be monitored for a follow-up period of 28 days. The findings of this study will be used to guide the Ministry of Health in evaluating its national policy for P. falciparum malaria treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 1 year
* Axillary temperature ≥ 37.5ºC and/or history of fever in the previous 48 hours without any other evident cause
* Unmixed infection with P. falciparum of between 250 and 100,000 asexual parasites/mm3 as determined by microscopic exam of the thick or thin smear
* An informed consent obtained from the patient or his/her guardian (in case of patients ≤ 18 years old) and assent for children (8-18 years old)
* Willingness to come to the health facility for the following 28 days

Exclusion Criteria:

* Signs or symptoms of severe malaria
* Other severe chronic diseases (e.g., cardiologic, renal, or hepatic diseases; HIV/AIDS; severe malnutrition)
* History of allergy to any of the proposed treatment or its alternatives, i.e. mefloquine, artesunate, quinine, tetracycline, or clindamycin
* Pregnancy (based on urine test), since this group of patients receives other drugs for malaria treatment in accordance with Peruvian national guidelines.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2005-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Macedo de Oliveira, MD, MSc, Principal Investigator — Centers for Disease Control and Prevention; Wilmer Marquiño Quezada, MD, Principal Investigator — National Institute of Health, Peru
Locations (1):
- Loreto Healthcare Facility, Iquitos, Loreto, Peru